CLINICAL TRIAL: NCT02530320
Title: Phase II Pilot, Prospective, Open Label, Multicenter CT, to Evaluate the Safety and Efficacy of Palbociclib (PD0332991), a Cyclin-dependent Kinase 4 and 6 (CDK4 and CDK6) Inhibitor, in Patients With Oligodendroglioma or Recurrent Oligoastrocytoma Anaplastic With the Activity of the Protein RB Preserved
Brief Title: Safety and Efficacy of PD0332991 (Palbociclib), a Cyclin-dependent Kinase 4 and 6 Inhibitor, in Patients With Oligodendroglioma or Recurrent Oligoastrocytoma Anaplastic With the Activity of the Protein RB Preserved
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Investigación en Neurooncología (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEINO 13
Record Dates: First submitted 2015-08-18; First posted 2015-08-21 (Estimated); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-10

CONDITIONS: Oligodendroglioma; Oligoastrocytoma
Keywords: Palbociclib; oligodendroglioma; oligoastrocytoma anaplastic
MeSH Terms: conditions — Oligodendroglioma; Astrocytoma | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Palbociclib (PD0332991) (Experimental): Palbociclib will be administrated orally at a dose of 125 mg/day during 21 days followed by a break of 7 days. All patients included will be treated in the same arm. Treatment will be administrated until disease progression, unacceptable adverse side effects or study end.
  Interventions: Drug: Palbociclib

INTERVENTIONS:
Drug: Palbociclib — Palbociclib will be administered orally at a dose of 125 mg/day, until disease progression, unacceptable adverse side effects or study end.
  Other Names: PD0332991

SUMMARY:
This multicenter, open-label, phase II trial aims to assess the safety and efficacy of palbociclib in adult patients with Oligodendroglioma or recurrent oligoastrocytoma anaplastic with the activity of the protein RB preserved.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and sign the informed consent approved by the Ethic Committee.
2. Men or women aged greater than or equal to 18.
3. Patients with oligodendroglioma anaplastic or oligoastrocytoma anaplastic according to WHO classification and histologically confirmed. Note: It can be included patients with oligoastrocytoma or oligodendroglioma G2 only if they have suffered a recurrence in which the diagnosis of the resection were G3.
4. Patients in relapse after radiotherapy and one or two lines of chemotherapy. Note: Both previous radiotherapy and chemotherapy could be received in adjuvant therapy or previous recurrences. It is also accepted to be received concurrent chemoradiotherapy. In the secondary oligodendrogliomas or oligoastrocytomas anaplastic, the patients could have received chemotherapy and radiotherapy when the tumor was G2.
5. All patients have to present positivity in immunohistochemical study for the RB protein in the tumor samples sent to the central lab.
6. The cases must have 10 slides or a tumor block available from a biopsy or surgery.
7. All patients have to show disease progression in a cerebral nuclear magnetic resonance.
8. Interval of at least one week between the previous intracranial biopsy and the inclusion.
9. Interval of at least 12 weeks between radiotherapy and the inclusion, unless: a) Recurrent tumor confirmed histologically b) recurrency showed in the NMR out of radiotherapy.
10. Patients should have been recovered from previous therapies: 28 days since the end of any investigational product and since the end of any cytotoxic treatment.
11. ECOG≤2
12. Stable or decreasing dose of corticoids during the five days prior to the inclusion
13. patients who have been suffered from a tumor resection in the last recurrence are eligible if:

    * A good surgery recover
    * there is a measurable or evaluable disease after surgery
14. Good bone marrow function:

    * Neutrophils ≥ 1500/mm3 (1.5x10e9/L)
    * Platelet ≥ 100.000/mm3 (100 x 10e9)
    * Hemoglobin ≥ 9 g/dL
    * Seric creatinine ≤ 1.5 x LSN of the site or estimated clearance ≥ 60 ml/min calculated.
    * Bilirubin ≤ 1.5 x LSN (if Gilbert's syndrome ≤ 3 xLSN) AST (SGOT) and/or ALT ≤ 3 x LSN; alkaline phosphatase ≤ 2.5 x LSN.
15. Nor pregnant women nor breast-feeding women. Women with heterosexual activity should have a negative pregnant test before the inclusion in the study. Both women and men should use an accepted contraceptive method during the study treatment and 1 month after treatment completed.

Exclusion Criteria:

1. Presence of meningeal carcinomatosis disseminated.
2. Concomitant treatment with other investigational products
3. Previous treatment wih an investigational product that could be active for CDK4/6
4. Any kind of surgery in the previous 2 weeks
5. Presence of any clinically significant gastrointestinal abnormality that can affect oral administration, transit or absorption of study drug, such as the inability to take medication by mouth as tablets.
6. Presence of any psychiatric or cognitive disorder that limits the understanding or the signature of informed consent and / or jeopardize the fulfillment of the requirements of this protocol.
7. In the 7 days prior to the beginning of the treatment, to have received a treatment with: - Drugs inhibitor of the CYP3A4 - Drugs inductors of the CYP3A4 - Drugs that extends the QT interval
8. QTc interval >480 msec, familiar history or personal of QT large Syndrome, QT short Syndrome, Brugada syndrome, QTc extension or Torsade de Pointes history
9. Electrolyte disorder that may affect the QTc interval
10. Significant or uncontrolled cardiovascular disease, including:

    * Myocardial infarction within the previous 12 months
    * Uncontrolled angina within the previous 6 months
    * Congestive heart failure in the previous 6 months
    * History of clinically significant ventricular arrhythmias of any type (as ventricular tachycardia, ventricular fibrillation or torsades de pointes)
    * History of second or third grade heart block (these patients may be eligible if you currently have a pacemaker)
    * Ictus
    * Pulmonary embolism
11. History of any cancer, except for the following circumstances:

    * Patients with a history of other malignancies are eligible if they have been free of disease for at least the last 3 years, and at the discretion of the investigator, there is low risk of disease recurrence.
    * Patients with the following cancers are eligible even if they are diagnosed and treated in the last 3 years: carcinoma in situ of the cervix and basal cell or basal cell skin carcinoma. Patients are ineligible if there is evidence of any neoplastic disease that required therapy other than surgery in the past 3 years.
12. Patients positive for HIV
13. Inflammatory bowel disease, chronic diarrhea, short gut syndrome or any upper gastrointestinal surgery including gastric resection.
14. History of allergic reactions to Palbociclib
15. Another acute or chronic serious medical condition, uncontrolled intercurrent illness or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of test results and that,investigator's discretion, make the patient inappropriate for entry into this trial. Uncontrolled intercurrent illness including, but are not limited to, ongoing or active infection or psychiatric illness / social situations that limit the compliance of study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-10-25 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Manuel Sepúlveda, Principal Investigator — H. 12 de Octubre
Locations (11):
- Spain (11):
  - Hospital Insular de Canarias, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Son Espases, Palma de Mallorca, Mallorca
  - Consorcio Hospitalario Provincial de Castellón, Castellon, Valencia
  - Hospital Clínic de Barcelona, Barcelona
  - ICO Hospitalet, Barcelona
  - Hospital de León, León
  - Hospital 12 de Octubre, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Regional de Málaga, Málaga
  - Hospital Virgen del Rocio, Seville
  - Hospital Universitario y Politécnico La Fe, Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 79 patients were screened and eventually 34 patients fulfilled all the inclusion and exclusion criteria.
Period: Overall Study
Arm/Group | Palbociclib (PD0332991)
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients With Recurrent Anaplastic (Grade III) Oligodendrogliomas.: All patients included in the study received treatment with the experimental drug, Palbociclib, at a dose of 125 mg/day on days 1-21 in 28-day cycles. The IMP was administered for 21 days followed by 7 days off. Treatment cycles continued until there was unacceptable toxicity, tumor progression, withdrawal of consent or death.
Arm/Group | Patients With Recurrent Anaplastic (Grade III) Oligodendrogliomas.
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: years] | 50.7 [30.7 to 68.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
ECOG, Categorical [Count of Participants; unit: Participants] — The ECOG-PS scale describes a patient's level of functioning in terms of their ability to care for them selves, and carry activities of daily living. The scale values are:
  0: Fully active, without restriction
  1. Restricted in physically strenuous activity but ambulatory
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Death
  Participants
    ECOG 0 | 10
    ECOG 1 | 19
    ECOG 2 | 5
Prior treatment Temozolomide [Count of Participants; unit: Participants]
  Temozolamide | 30
  Nitrosoureas | 23
  Radiotherapy | 34

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) at Six Months (PFS6m)
Description: Percentage of patients who have progressed / no progress after 6 months of treatment
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Patients With Recurrent Anaplastic (Grade III) Oligodendrogliomas.: Patients with recurrent anaplastic (Grade III) oligodendrogliomas ith preservation of activity of the RB protein.
Arm/Group | Patients With Recurrent Anaplastic (Grade III) Oligodendrogliomas.
Number analyzed (Participants) | 34
Percentage of participants | 21 [11 to 41]

2. Secondary Outcome: Safety and Tolerability of Oral Administration of PD0332991 (Reported Adverse Events, Physical Examinations and Laboratory Tests. Toxicity Will be Classified and Tabulated by NCI-CTCAE v 4.0.)
Description: Type, incidence, severity, frequency, severity and relationship with IMP of reported adverse events, physical examinations and laboratory tests. Toxicity will be classified and tabulated by NCI-CTCAE v 4.0.
Time Frame: Three years
Population: Palbociclib will be administrated orally at a dose of 125 mg/day during 21 days followed by a break of 7 days. All patients included will be treated in the same arm. Treatment will be administrated until disease progression, unacceptable adverse side effects or study end.
  Palbociclib: Palbociclib will be administered orally at a dose of 125 mg/day, until disease progression, unacceptable adverse side effects or study end.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib (PD0332991)
Number analyzed (Participants) | 34
Participants
  Adverse envents (any) | 33
  Adverse events (≥ Grade 3) | 25
  TRAEs (any) | 29
  TRAEs (≥ Grade 3) | 22
  SAE (any) | 7
  SAE no related | 7
  Toxicity (any) | 29
  Toxicity grade≥3 | 22

3. Secondary Outcome: Anti-tumor Response According to RANO Criteria
Description: According to RANO criteria, assessed by the PI of each center. There will be a central review.
Time Frame: 30 months
Population: Patients with recurrent anaplastic (Grade III) oligodendrogliomas
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Recurrent Anaplastic (Grade III) Oligodendrogliomas.
Number analyzed (Participants) | 34
Participants
  No evaluated | 1
  Stable disease (SD) | 13
  Progression disease (PD) | 20

4. Secondary Outcome: Overall Survival (OS)
Description: Time from randomization to death by any cause.
Time Frame: With a median follow-up of 12 (0.9-52.2) months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Patients With Recurrent Anaplastic (Grade III) Oligodendrogliomas.
Number analyzed (Participants) | 34
months | 32 [11 to NA] — upper limit of confidence interval not estimable due to an insufficient number of participants with events

5. Secondary Outcome: Changes in the Use of Glucocorticoids
Description: Percentage of patients decreasing doses of corticosteroids during treatment. Corticoids evolution
Time Frame: 30 months
Population: Percentage of patients decreasing doses of corticosteroids during treatment. Corticoids evolution
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Recurrent Anaplastic (Grade III) Oligodendrogliomas.
Number analyzed (Participants) | 34
Participants
  NA or not reported | 7
  Decrease | 1
  Increase | 3
  No corticoids | 21
  Stable | 2

ADVERSE EVENTS:
Time Frame: Adverse events will be monitored from first dose of study treatment until 30+/-3 days after end of treatment, an average of three years Events will be followed up until resolved or deemed irreversible, which what happens later.
Arm/Group | Patients With Recurrent Anaplastic (Grade III) Oligodendrogliomas.
All-Cause Mortality (participants affected / at risk) | 16/34
Serious Adverse Events (participants affected / at risk) | 7/34
Other Adverse Events (participants affected / at risk) | 24/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Recurrent Anaplastic (Grade III) Oligodendrogliomas. (N=34)
Ataxia - G2 (Nervous system disorders) | 1 (1) — No relation; Intensity: Hospitalization; Action: None
Cognitive disturbance - G3 (General disorders) | 1 (1) — No relation; Intensity: Hospitalization; Action: Delay of treatment
Seizure - G2 (General disorders) | 1 (1) — Relation:No; Intensity: Hospitalization; Action: None
Dysphasia - G3 (General disorders) | 1 (1) — Relation: No; Intensity: Hospitalization; Action: None
Surgical and medical procedures - Other, glioma exeresis - G1 (Surgical and medical procedures) | 1 (1) — No Relation; Intensity: Relevant medical; Action:None
Cognitive impairment - G3 (General disorders) | 1 (1) — Relation: No; Intensity: Hospitalization; Action: None
General disorders and administration site conditions - Other, clinical deterioration - G3 (General disorders) | 1 (1) — Relation: No; Intensity: Hospitalization; Action: None
Hyperglycaemia - G4 (Metabolism and nutrition disorders) | 1 (1) — Relation: No; Intensity: Hospitalization; Action:None
Confusion - G3 (General disorders) | 1 (1) — Relation:No; Intensity: Hospitalization; Interruption of treatment
Muscle weakness left-sided - G2 (Musculoskeletal and connective tissue disorders) | 1 (1) — Relation: No Intensity: Hospitalization. Action: None
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Recurrent Anaplastic (Grade III) Oligodendrogliomas. (N=34)
Neutrophil count decreased (Immune system disorders) | 24 (24)
Fatigue (Respiratory, thoracic and mediastinal disorders) | 20 (20)
Platelet count decreased (Blood and lymphatic system disorders) | 17 (17)
Anaemia (Blood and lymphatic system disorders) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 6 (6)
Cognitive disturbance (Nervous system disorders) | 5 (5)
Seizure (Nervous system disorders) | 4 (4)
Flu like symptoms (General disorders) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 5 (5)
Cephalea (Nervous system disorders) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (3)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 3 (3)
Fever (General disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3)
Confusion (Psychiatric disorders) | 2 (2)
Cognitive impairment (Nervous system disorders) | 2 (2)
White blood cell decreased (Blood and lymphatic system disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Injury, poisoning and procedural complications - other, Lip wound (Injury, poisoning and procedural complications) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT02530320/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/20/NCT02530320/SAP_001.pdf